CLINICAL TRIAL: NCT05511116
Title: Neoadjuvant Treatment of Resectable or Locally Advanced Borderline Pancreatic Adenocarcinoma: Reproducibility of Tumor Measurement in CT Versus MRI
Brief Title: Neoadjuvant Treatment of Resectable or Locally Advanced Borderline Pancreatic Adenocarcinoma: Reproducibility of Tumor Measurement in CT VS MRI
Acronym: ReMeTTI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ReMeTTI
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Pancreas Cancer; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite important therapeutic advances, pancreatic adenocarcinoma remains one of the cancers with a high mortality rate (4th leading cause of cancer death in the US in 2021), poor prognosis (5-year overall survival rate of 10%) and increasing incidence.

Patients are often metastatic from the start or at an advanced stage at diagnosis, making curative treatment difficult to envisage. Although the gold standard of treatment for resecable pancreatic adenocarcinoma is initial surgery followed by adjuvant chemotherapy, considerable interest has emerged in a treatment strategy involving neoadjuvant therapy in patients at high risk for positive resection margins (R1) on initial imaging workup.

The assessment of response to neoadjuvant therapy is complex, especially for the evaluation of vascular invasion with a high risk of overestimating residual invasion after neoadjuvant therapy. Accurate assessment of tumor size before and after neoadjuvant treatment is therefore crucial to identify good responders (according to RECIST 1.1 criteria) and thus improve the selection of patients who can benefit from curative surgery with healthy resection margins (R0).

In clinical practice, tumor size assessment is performed by injected computed tomography (CT). The latter has certain advantages in terms of technical reproducibility, but has a number of limitations. Indeed, the delineation of the tumor mass in CT seems to be subject to a significant inter-observer variability. The same is true for vascular invasion. CT also seems to underestimate the size of the tumor compared to the anatomopathological examination of the surgical specimen. On the other hand, Magnetic Resonance Imaging (MRI) has been shown to be superior to CT in tumor detectability and diagnosis of malignancy in the presence of an indeterminate pancreatic mass. It has also been shown that tumor size, whether measured in diameter or volume, is frequently underestimated on CT compared to multiparametric MRI or pathological examination of the resection specimen.

In the latest recommendations of the National Comprehensive Cancer Network (NCCN), MRI is indicated at diagnosis in non-metastatic patients with indeterminate liver lesions on CT, or as a second-line alternative to CT for re-evaluation after neo-adjuvant therapy in patients with resectable or borderline resectable disease according to the NCCN classification. However, MRI is increasingly performed routinely in some centers, both at diagnosis and at re-evaluation after neo-adjuvant therapy. The question of which imaging modality between CT and multiparametric MRI is the most reproducible in terms of tumor size measurement becomes important, especially in the evaluation of the response to neoadjuvant therapy. A few studies have investigated the interobserver variability of tumor size measurement in CT versus MRI in the context of radiotherapy management for the delineation of an irradiation field, but to date investigators have not found any study evaluating the interobserver variability of tumor size measurement using RECIST criteria before and after neoadjuvant treatment for pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with histologically proven pancreatic adenocarcinoma (biopsy or resection specimen)
* Non-metastatic (M0) on the PCR form
* Patient who received chemotherapy or radio-chemotherapy first
* MRI and CT scans performed before or at the beginning of neo-adjuvant (or induction) treatment, during treatment and/or at the end of neo-adjuvant treatment (but before excision surgery)
* French-speaking patient

Exclusion Criteria:

* Patients who object to the use of their data for this research
* Patients operated on immediately without neoadjuvant treatment
* Patients for whom re-evaluation MRI or CT is not available or has not been done
* Patients for whom the re-evaluation MRI or CT scan was performed more than 60 days before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven pancreatic adenocarcinoma (biopsy or resection specimen), Non-metastatic (M0) on the PCR form, whom received chemotherapy or radio-chemotherapy first.
  MRI and CT scans performed before or at the beginning of neo-adjuvant (or induction) treatment, during treatment and/or at the end of neo-adjuvant treatment (but before excision surgery).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Inter-observer reproducibility | Month 3
  This outcome corresponds to the comparison of tumor measurements of pancreatic adenocarcinomas between the 3 readers for each examination (MRI and CT).

SECONDARY OUTCOMES:
Performances de la mesure tumorale par TDM vs. IRM | Month 3
  This outcome corresponds to the diagnostic performance of CT vs. MRI with reference to pathological examination.
Tumor response on morphological imaging vs. tumor response grade on pathology | Month 3
  This outcome corresponds to the Comparison of pathological FIT to morphological response by CT vs. MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Marc ZINS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Saad AM, Turk T, Al-Husseini MJ, Abdel-Rahman O. Trends in pancreatic adenocarcinoma incidence and mortality in the United States in the last four decades; a SEER-based study. BMC Cancer. 2018 Jun 25;18(1):688. doi: 10.1186/s12885-018-4610-4. PMID 29940910
- [Background] Kaufmann B, Hartmann D, D'Haese JG, Stupakov P, Radenkovic D, Gloor B, Friess H. Neoadjuvant Treatment for Borderline Resectable Pancreatic Ductal Adenocarcinoma. Dig Surg. 2019;36(6):455-461. doi: 10.1159/000493466. Epub 2018 Nov 8. PMID 30408790
- [Background] Tempero MA, Malafa MP, Al-Hawary M, Behrman SW, Benson AB, Cardin DB, Chiorean EG, Chung V, Czito B, Del Chiaro M, Dillhoff M, Donahue TR, Dotan E, Ferrone CR, Fountzilas C, Hardacre J, Hawkins WG, Klute K, Ko AH, Kunstman JW, LoConte N, Lowy AM, Moravek C, Nakakura EK, Narang AK, Obando J, Polanco PM, Reddy S, Reyngold M, Scaife C, Shen J, Vollmer C, Wolff RA, Wolpin BM, Lynn B, George GV. Pancreatic Adenocarcinoma, Version 2.2021, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2021 Apr 1;19(4):439-457. doi: 10.6004/jnccn.2021.0017. PMID 33845462
- [Background] Soloff EV, Al-Hawary MM, Desser TS, Fishman EK, Minter RM, Zins M. Imaging Assessment of Pancreatic Cancer Resectability After Neoadjuvant Therapy: AJR Expert Panel Narrative Review. AJR Am J Roentgenol. 2022 Apr;218(4):570-581. doi: 10.2214/AJR.21.26931. Epub 2021 Dec 1. PMID 34851713
- [Background] Dalah E, Moraru I, Paulson E, Erickson B, Li XA. Variability of target and normal structure delineation using multimodality imaging for radiation therapy of pancreatic cancer. Int J Radiat Oncol Biol Phys. 2014 Jul 1;89(3):633-40. doi: 10.1016/j.ijrobp.2014.02.035. Epub 2014 Apr 20. PMID 24755533
- [Background] Legrand L, Duchatelle V, Molinie V, Boulay-Coletta I, Sibileau E, Zins M. Pancreatic adenocarcinoma: MRI conspicuity and pathologic correlations. Abdom Imaging. 2015 Jan;40(1):85-94. doi: 10.1007/s00261-014-0196-8. PMID 25030776